CLINICAL TRIAL: NCT06595784
Title: The HELlenic Thoracic Society Initiative for CΟPD and CVD
Acronym: HELICOPD
Status: Recruiting | Type: Observational
Sponsor: Hellenic Thoracic Society (Other)
Responsible Party: Sponsor
Other Study IDs: HTS001
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Cardiovascular Diseases (CVD)
Keywords: Chronic obstructive pulmonary disease; COPD; Cardiovascular disease; CVD; Protocol; Real-World Data
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COPD patients with cardiovascular comorbidities

SUMMARY:
COPD is one of the most common respiratory diseases in Greece, and maybe more than half a million Greek citizens suffer both from COPD and CVD, however their characteristics and management remain unknown. HELICOPD is a national, multicenter, prospective, non-interventional study designed to contribute to better understanding and depicting the demographic and clinical characteristics of this population, the COPD- and CVD-related adverse events in a two-years period, their quality of life and the healthcare resources use. The study is initiated and coordinated by the Hellenic Thoracic Society.

ELIGIBILITY:
Inclusion criteria

Patients should cumulatively meet the following three (3) criteria to be enrolled in the study:

1. To have been diagnosed with chronic obstructive pulmonary disease and at least one cardiovascular comorbidity (heart failure, atherosclerotic cardiovascular disease, atrial Fibrillation, severe valvular disease)
2. Adults aged >35 years at the time of inclusion in the study,
3. With signed informed consent for their participation in the study. Exclusion criteria Patients with the below limitations are not eligible to participate in the study

Patients:

1. Without at least one cardiovascular comorbidity,
2. With history of lung cancer
3. With any other active malignancy and undergoing treatment (chemotherapy/radiotherapy/immunotherapy)
4. With any thoracic or abdominal surgery planned during study follow-up period
5. With participation in any COPD-related interventional study at study entry or during study duration.
6. Without signed informed consent for their participation in the study.

Ages: 35 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD and cardiovascular comorbidities in Greece
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of moderate or severe COPD exacerbations | Up to 24 months
  Moderate COPD exacerbation: typically requires outpatient management, it is characterized by an increased need for medication, specifically the use of systemic corticosteroids and/or antibiotics. Severe COPD exacerbation: indicated by an acute worsening of symptoms that requires hospitalization.
Number of cardiovascular complications/outcomes | Up to 24 months
  Cardiovascular complications/outcomes, including a) acute coronary syndrome, b) ischemic stroke, c) pulmonary embolism, d) reperfusion, e) worsening of heart failure that required a visit to the Emergency Department (ED) or hospitalization (short or longer), f) other hospitalization in a cardiology clinic (causes other than acute coronary syndrome, reperfusion, and heart failure), g) death related to cardiovascular disease.

SECONDARY OUTCOMES:
Unscheduled hospital admission due to COPD | Up to 24 months
Unscheduled hospital admission due to any other reason | Up to 24 months

OTHER OUTCOMES:
Death (due to any cause) | Up to 24 months
Healthcare resource utilization related costs | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Hillas, Principal Investigator — 5th Pulmonary Department, "Sotiria" Chest Diseases Hospital, Athens, Greece; Paschalis Steiropoulos, Principal Investigator — Department of Respiratory Medicine, Medical School, Democritus University of Thrace, University General Hospital
Locations (2):
- Greece (2):
  - Department of Respiratory Medicine, Medical School, Democritus University of Thrace, University General Hospital, Alexandroupoli
  - 5th Pulmonary Department, "Sotiria" Chest Diseases Hospital, Athens, Greece, Athens